CLINICAL TRIAL: NCT05353478
Title: Reducing Opioids After Percutaneous Stone Surgery
Brief Title: Reducing Opioid Prescription After Kidney Stone Removal Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kevin Koo, Principal Investigator, Mayo Clinic
Other Study IDs: 22-000494
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Kidney Stone
Keywords: Percutaneous Nephrolithotomy (PCNL)
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to implement and assess a standard way of prescribing opioid pain medication following PCNL (a kidney stone removal surgery) to ensure patients are being discharged with an appropriate quantity of pain management medication.

DETAILED DESCRIPTION:
Participants in this study will have their opioid pain medication prescription at discharge following PCNL (Percutaneous Nephrolithotomy, a kidney stone removal surgery) determined by an algorithm in addition to physician judgement. The goal of the algorithm is help physicians refine pain medication prescribing patterns for patients who have undergone PCNL in order to discharge patients with an appropriate quantity of pain management medication. The effectiveness of the algorithm will be assessed through participant surveys. Participants will complete a brief online survey on Days 3, 7, and 14 following hospital discharge and another phone-based survey 26-30 days after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing percutaneous nephrolithotomy at Mayo Clinic Rochester.

Exclusion Criteria:

* Unable or unwilling to provide informed consent.
* Patients who require Intensive Care Unit admission after surgery.
* Patients who have Clavien grade III or greater postoperative complications requiring additional intervention < 30 days after index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing percutaneous nephrolithotomy at Mayo Clinic Rochester.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Unused opioid prescriptions | 30 days
  Number of unused opioids following recovery from percutaneous nephrolithotomy

SECONDARY OUTCOMES:
Unfilled opioid prescriptions | 30 days
  Number of unfilled opioid prescriptions following recovery from percutaneous nephrolithotomy
Opioid prescription refills | 30 days
  Number of opioid prescription refills following recovery from percutaneous nephrolithotomy

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Koo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials